CLINICAL TRIAL: NCT03491904
Title: A Phase 1, Multicenter, Randomized, Open-Label, Parallel-Group, Multi-Dose Study in Patients With Moderate-to-Severe Pain Due to Osteoarthritis of the Knee or Hip to Assess the Patients' Ability to Self-Administer Fasinumab Using an Auto-Injector and to Characterize the Pharmacokinetics of Fasinumab Using Two Different Presentations
Brief Title: To Assess the Patients' Ability to Self-Administer Fasinumab
Acronym: FACT DEVICE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R475-PN-1602
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — fasinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Auto-injector (AI) (Experimental)
  Interventions: Drug: Fasinumab AI
- Prefilled syringe (PFS) (Experimental)
  Interventions: Drug: Fasinumab PFS

INTERVENTIONS:
Drug: Fasinumab AI — Self-administered with auto injector
  Other Names: REGN475
  Arms: Auto-injector (AI)
Drug: Fasinumab PFS — Prefilled syringe administered by study staff
  Other Names: REGN475
  Arms: Prefilled syringe (PFS)

SUMMARY:
The primary objective is to demonstrate that the auto-injector(AI) is suitable to be used to administer fasinumab at home by patients or their caregivers, as measured by collecting 12 weeks of actual-use data on the technical performance of the device.

The secondary objectives of the study are:

* To evaluate the successful injection of fasinumab by patients or their caregivers using the AI in an unsupervised setting
* To evaluate patient/caregiver satisfaction with the AI for fasinumab injection in an unsupervised setting
* To evaluate exposure in serum for fasinumab administered by patients or their caregivers using an AI in an unsupervised setting, or fasinumab administered by study staff using a PFS that has been used in the phase 3 program
* To characterize the safety, tolerability, and immunogenicity of fasinumab administered by patients or their caregivers using an AI in an unsupervised setting, or fasinumab administered by study staff using a PFS that has been used in the phase 3 program

ELIGIBILITY:
Key Inclusion Criteria:

1. A clinical diagnosis of Osteoarthritis (OA) of the knee or hip based on the American College of Rheumatology criteria with radiologic evidence of OA (K-L score ≥2 for the index joint) at the screening visit
2. Moderate-to-severe pain in the index joint defined as a WOMAC average pain subscale score of ≥4 at both the screening and randomization visits
3. Willing to discontinue current pain medications and to adhere to study requirements for rescue treatments
4. A history of at least 12 weeks of analgesic use for pain due to OA of the knee or hip
5. History of regular use of analgesic medications for OA pain (defined as an average of 4 days per week over the 4 weeks prior to the screening visit), including NSAIDs, selective cyclooxygenase 2 inhibitors, opioids, paracetamol/acetaminophen, or combinations thereof

Key Exclusion Criteria:

1. History or presence at the screening visit of non-OA inflammatory joint disease (eg,rheumatoid arthritis, lupus erythematosus, psoriatic arthritis, pseudo-gout, gout, spondyloarthropathy, polymyalgia rheumatica, joint infections within the past 5 years), Paget's disease of the spine, pelvis or femur, neuropathic disorders, multiple sclerosis, fibromyalgia, tumors or infections of the spinal cord, or renal osteodystrophy
2. History or presence on imaging of arthropathy (osteonecrosis, subchondral insufficiency fracture, rapidly progressive OA type 1 or type 2), stress fracture, recent stress fracture, neuropathic joint arthropathy, hip dislocation (prosthetic hip dislocation is eligible), knee dislocation (patella dislocation is eligible), congenital hip dysplasia with degenerative joint disease, extensive subchondral cysts, evidence of bone fragmentation of collapse, or primary metastatic tumor with the exception of chondromas or pathologic fractures during the screening period
3. Trauma to the index joint within 3 months prior to the screening visit
4. Signs or symptoms of carpal tunnel syndrome within 6 months of screening
5. Patient is not a candidate for MRI

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Percentage of device-associated product technical failure (PTF) for the AI based on the total number of fasinumab injections administered by patients/caregivers in an unsupervised setting | Baseline to Week 16

SECONDARY OUTCOMES:
Proportion of successful fasinumab injections administered by patients or their caregivers using an AI in an unsupervised setting (per patient report) | Baseline to Week 16
Number of AI associated product technical complaint (PTCs) | Baseline to Week 16
Number of validated AI associated PTFs | Baseline to Week 16
Number of patients with an AI associated PTC | Baseline to Week 16
Number of AI use-related errors | Baseline to Week 16
  Including but not limited to improper storage, inappropriate use of the device, dosing schedule mistakes, and user handling mistakes
Patient satisfaction with the AI as assessed using the Self-Injection Assessment Questionnaire (SIAQ) | Baseline to Week 16
Number of participants who experience Adjudicated arthropathy (AA) | Through week 36
  As confirmed by independent adjudication
Number of participants who experience Destructive arthropathy (DA) | Through week 36
  As confirmed by independent adjudication
Number of participants who experience treatment-emergent adverse events (TEAEs) | Through week 16
Number of participants who experience sympathetic nervous system dysfunction | Through week 36
Number of participants who experience peripheral sensory adverse events (AEs) that require a neurology or other specialty consultation | Through week 36
Number of participants who experience all-cause Joint replacement (JR)s | Through week 36
Number of participants who experienced JR at the telephone survey | 52 weeks after last dose of study drug
Maximum observed drug concentration (Cmax) | Up to 36 weeks
Area under the curve from the time of dosing to the end of dosing interval (AUC) | Up to 36 weeks
Geometric mean ratio of Cmax and AUC for the AI device (CI) of the geometric mean ratio | Up to 36 weeks
Geometric mean ratio of Cmax and AUC for the PFS device (CI) of the geometric mean ratio | Up to 36 weeks
Incidence of anti-drug antibody (ADA) | Up to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (20):
- United States (20):
  - Regeneron Research Facility, Gilbert, Arizona
  - Regeneron Research Facility, Glendale, Arizona
  - Regeneron Research Facility, Los Angeles, California
  - Regeneron Research Facility, Wheat Ridge, Colorado
  - Regeneron Research Facility, Ocala, Florida
  - Regeneron Research Facility, Orlando, Florida
  - Regeneron Research Facility, Pinellas Park, Florida
  - Regeneron Research Facility, Port Orange, Florida
  - Regeneron Research Facility, Atlanta, Georgia
  - Regeneron Research Facility, West Des Moines, Iowa
  - Regeneron Research Facility, Wichita, Kansas
  - Regeneron Research Facility, Lexington, Kentucky
  - Regeneron Research Facility, Jamaica, New York
  - Regeneron Research Facility, Statesville, North Carolina
  - Regeneron Research Facility, Wilmington, North Carolina
  - Regeneron Research Facility, Oklahoma City, Oklahoma
  - Regeneron Research Facility, Bristol, Tennessee
  - Regeneron Research Facility, Knoxville, Tennessee
  - Regeneron Research Facility, Dallas, Texas
  - Regeneron Research Facility, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual de-identified participant data will be made available once the indication has been approved by a regulatory body, if there is participant consent and there is not a reasonable likelihood of participant re-identification
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/